CLINICAL TRIAL: NCT06673459
Title: Busulfan Plus Cyclophosphamide Vs. Total Body Irradiation Plus Cyclophosphamide for Allogeneic Hematopoietic Stem Cell Transplantation in Patients with Acute T Lymphoblastic Leukemia: a Randomized Controlled, Open-label, Multi-center Clinical Trial
Brief Title: BuCy Vs. TBICy for Allo-HSCT in T-ALL Patients
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Children's Hospital of Soochow University (Other); Ruijin Hospital (Other); Nanfang Hospital, Southern Medical University (Other); Fujian Medical University Union Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Zhejiang University (Other); Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Yang Xu, The First Affiliated Hospital of Soochow University, The First Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TREAL1
Record Dates: First submitted 2024-11-02; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-05

CONDITIONS: T-Cell Lymphocytic Leukemia; ALLOGENEIC HEMATOPOIETIC STEM CELL TRANSPLANTATION; Total Body Irradiation; Chemotherapy
MeSH Terms: conditions — Leukemia, T-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TBICy (Experimental): Patients enrolled in this arm will receive total body irradiation plus cyclophosphamide as conditioning regimen.
  Interventions: Biological: TBICy
- BuCy (Active Comparator): Patients enrolled in this arm will receive busulfan plus cyclophosphamide as conditioning regimen.
  Interventions: Biological: BuCy

INTERVENTIONS:
Biological: TBICy — The TBI-Cy group was administered 250 mg/m2/d oral Me-CCNU on day -8. A total of 12 Gy TBI was for each patient and fractionated dose was 2 Gy twice daily or 4Gy once daily on days -8 to -6. Occluding of the lung fields during TBI, the corresponding irradiation dose reduced to a total of 8 Gy. On day -5, the schedule was intravenous 2 g/m2 Ara-C every 12 hours. Then intravenous 1.8 g/m2 CTX once per day from days -4 to -3.
  Arms: TBICy
Biological: BuCy — The BuCy group received oral Me-CCNU 250 mg/m2/d twice daily on day -8, intravenous cytosine arabinoside (Ara-C) 2 g/m2 twice daily on day -7, intravenous Bu 3.2 mg/kg/d from days -6 to -4, and intravenous cyclophosphamide (CTX) 1.8 g/m2/d from days -3 to -2. There were no patients accepted oral Bu.
  Arms: BuCy

SUMMARY:
T-cell acute lymphoblastic leukemia (T-ALL), a hematological malignant neoplasm of immature T cells, accounting for a morbidity of 10-15% among pediatric and 20-25% among adult patients of ALL. Despite the application of improved intensive therapies, the overall survival (OS) of T-ALL patients is still unsatisfactory, with a 5-year OS rate of less than 60% in adults and 85% in children. Over the past few decades, allogeneic hematopoietic stem-cell transplantation (allo-HSCT) has emerged as a potential and the most likely curative treatment for patients with high-risk hematological malignant neoplasms, and it has been proven that allo-HSCT could hold the potential to improve the prognosis of T-ALL patients and may even cure T-ALL.

The two most common myeloablative conditioning regimens for T-ALL patients with allo-HSCT were total body irradiation (TBI) plus cyclophosphamide (TBI-Cy) and busulfan (Bu) plus cyclophosphamide (BuCy). The most common use conditioning regimen for ALL patients is the TBI-Cy conditioning regimen over other hematological malignancy patients because TBI possess potent and distinct anti-leukemic effects, particularly in organs not easily affected by systemic chemotherapy and intense immunosuppressive effects. However, TBI-based conditioning regimens may cause a high risk of cataracts, interstitial pneumonitis (IP), engraftment failure and even subsequent malignant neoplasms (SMNs). To avoid these disadvantages, intravenous Bu replaced TBI as a part of conditioning.

Extensive studies have shown that allo-HSCT with conditioning regimens based on TBI could benefit survival compared with conditioning regimens based on chemotheraphy in treating ALL. We retrospectively analyzed post-10-year data from T-ALL patients from two transplant centers, and all the databases were used to eliminate confounding factors via PSM. We demonstrated that the TBI-Cy conditioning regimen had inferior efficacy to the BuCy conditioning regimen, especially for T-ALL patients who were children, refractory, had extramedullary disease before transplantation, had active disease or an MRD-positive status at allo-HSCT, or who received haplo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

1. T-ALL patients aged > 2 years and ≤55 years;
2. For the first time accept allo-HSCT;
3. With Eastern Cooperative Oncology Group (ECOG) performance status of 0-3; 4. Signing an informed consent form, having the ability to comply with study and follow-up procedures.

Exclusion Criteria:

1. With other malignancies;
2. With a previous history of autologous hematopoietic cell transplantation, allogeneic hematopoietic cell transplantation or chimeric antigen receptor T cell therapy;
3. With uncontrolled infection intolerant to haploidentical hematopoietic cell transplantation;
4. With severe organ dysfunction;
5. In pregnancy or lactation period;
6. With any conditions not suitable for the trial (investigators' decision).

Ages: 2 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 430 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2029-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2 years after randomization
  estimated progression-free survival at 2 year

SECONDARY OUTCOMES:
Overall survival | 2 years after randomization
  estimated overall survival at 2 year
Cumulative incidence of relapse | 2 years after randomization
  estimated cumulative incidence of relapse at 2 year
Non-relapse mortality | 2 years after randomization
  estimated non-relapse mortality at 2 year
Adverse events | 2 years after randomization
  Number of participants with adverse events. Frequencies of toxicities based on Common Terminology Criteria for Adverse Events (CTCAE) will be tabulated.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No